CLINICAL TRIAL: NCT03858127
Title: Preliminary Study on Activation of the Hypothalamic-pituitary-gonadal Axis in Infancy (Minipuberty) and Its Effects on Catch-up Growth and Neurocognitive Outcome in Male Preterm Neonates Born at <32 Weeks of Gestational Age
Brief Title: Minipuberty and Its Effects on Preterm Neonates
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Other Study IDs: GN18ME668P
Record Dates: First submitted 2019-02-15; First posted 2019-02-28 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-02

CONDITIONS: Infant, Newborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Male infants born <32 weeks gestation
  Interventions: Other: Collection of urine sample; Other: Examination of genitalia; Other: Video messaging

INTERVENTIONS:
Other: Collection of urine sample — Collection of urine sample for measurement of LH and FSH
Other: Examination of genitalia — Examination of genitalia
Other: Video messaging — Short video of infant recorded at home by the parents

SUMMARY:
It is generally known that there are some hormonal changes during puberty, but the knowledge about the activation of the same hormonal axis in the first months of life is relatively recent and it is not completely understood.

From the first weeks of life there is a progressive increase in hormone levels and this post-natal activation is called "minipuberty". Particularly in males, testosterone and androgen levels are associated with development and maturation of the reproductive system as well as changes in the brain structure and behaviours. Recently, it has also been suggested that the increasing testosterone level during the first 6 months of life, as well as during puberty, translates into an increase of linear growth.

In preterm neonates these hormones rise higher and for longer than in full-term newborns, suggesting that its activity is evolutionarily regulated.

With this study researchers would like to investigate these changes and correlate hormone levels with linear growth and neurobehavioral development of preterm infants.

DETAILED DESCRIPTION:
The activation of the hypothalamic-pituitary-gonadal axis (HPG) develops through three main moments: foetal life, first postnatal months (usually first 6 months of life) and finally during puberty. During the foetal period, there is a peak of gonadotropin secretion starting from the second trimester of gestation, and a subsequent suppression in the last weeks until birth, due to the negative feedback of placental estrogens. In male foetuses, LH levels exceed those of FSH. The foetal testis secretes testosterone and anti-müllerian hormone (AMH) from the 8th week of gestation and this is essential for masculinization. Formation of the active metabolite of testosterone, dihydrotestosterone, is required for the development of the prostate, penis and scrotum. Initial testicular development is intra-abdominal and the descent of the testes into the scrotum occurs in two phases. The first, transabdominal, phase is completed by 15 weeks of gestation. The second, inguinoscrotal, phase is usually completed by the end of the 35th week of gestation and this phase is androgen dependent. Testosterone levels are high in male foetuses between 10 and 20 weeks of gestational age, reaching adult values, and decrease thereafter towards term. In the same way LH and FSH levels decrease towards the end of gestation and are low at term in both sexes, due to the negative feedback of placental oestrogens.

A second post-natal HPG activation, also called "minipuberty", occurs at around 1 week of age, when placental hormones are cleared from the circulation. From the first weeks of life onwards there is a progressive increase in gonadotropins levels with a greater increase of FSH in females and of LH in males. During the "minipuberty" period gonadotropins levels have a peak at 3 months of life and a progressive exhaustion at around 6 months, except for FSH levels in females that can remain high even up to 3 or 4 years. Particularly in males, testosterone and androgen levels are associated with development and maturation of the reproductive system (penis and testis) as well as the androgynous cutaneous manifestations and a different neurobehavioral structure. Postnatal testosterone levels have been associated with male-type behaviour in 14-month-old infants, suggesting a role in neurobehavioral development.6 Recently, it has also been suggested how the increasing testosterone level during the first 6 months of life, as well as during puberty, translates into an increase of linear growth, regardless of the levels of growth hormone (GH) or insulin-like growth factor (IGF1).

Preterm birth does not seem to influence post-natal HPG activation, since that gonadotropin levels seem to raise up at the same time as term infants after the birth. The difference is that in preterm neonates these values last higher and longer than full-term newborns. According to the most recent longitudinal data, the post-natal activity of this axis declines at about the same in term neonates compared to premature infants with the same corrected gestational age, suggesting that the HPG activity is evolutionarily regulated. This higher increase of gonadotropin levels in premature males has been associated with a faster penile and testicular growth after birth compared to full-term boys. At last, in neonates small for gestational age (SGA) there are some evidence that post-natal FSH and testosterone levels are higher compared to infants with an adequate weight (AGA), although it is not known whether this correlates or have any influence on the catch-up growth of this subjects.

Understanding how "minipuberty" can influence linear growth, genitalia development and neurocognitive processes in preterm neonates has a significant scientific impact and could provide more information in understanding auxological and neurobehavioral developmental patterns of this population.

ELIGIBILITY:
Inclusion Criteria:

* Male preterm infants born ≤32 weeks of gestational age
* Written informed consent provided

Exclusion Criteria:

* Female sex assignment at birth
* Male preterm infants born >32 weeks of gestational age
* Male infants born at term

Max Age: 72 Hours | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Male infants
Study Population: We aim to enroll 20 neonates born under 32 weeks of gestational age at the Royal Hospital for Children in Glasgow. Neonates will be enrolled during the first 3 days of life with written informed consent signed by their parents.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Measurement of urinary luteinising hormone | 18 months
  Urinary LH measured every week on fresh samples using electro- chemiluminescence immunoassay (ECLIA). Sample analysis will be performed by the Biochemistry Department of the Royal Hospital for Children in Glasgow using Abbott Architect i1600 instrument
Measurement of urinary follicle stimulating hormone | 18 months
  Urinary FSH measured every week on fresh samples using electro- chemiluminescence immunoassay (ECLIA). Sample analysis will be performed by the Biochemistry Department of the Royal Hospital for Children in Glasgow using Abbott Architect i1600 instrument

SECONDARY OUTCOMES:
Measurement of weight | 18 months
  Each baby will have a naked weekly weight as part of their routine care, using calibrated weighing scales
Measurement of occipital frontal circumference | 18 months
  Each baby will have a weekly OFC measured as part of their routine care using a measuring tape
Measurement of penile growth | 18 months
  Each baby will have a weekly penile length measured using a measuring tape
Measurement of penile volume | 18 months
  Each baby will have penile volume measured weekly using an orchidometer
Video recording of fidgety movements | 18 months
  Each baby will have a 4-5 minute video recording taken by their parents for Prechtl's Method For The Qualitative Assessment Of General Movements

CONTACTS AND LOCATIONS:
Overall Officials: Paul Dearie, Study Director — NHS GGC R&D

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03858127/Prot_SAP_000.pdf